CLINICAL TRIAL: NCT06173089
Title: REmote MOnitoring of paTiEnts witH pacEmaker or implAntable cardioverteR defibrillaTor
Acronym: REMOTE-HEART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: 4279-1/2022
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
Keywords: remote monitoring; home monitoring; heart failure; cardiac resynchronization therapy; implantable cardioverter defibrillator
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Remote monitoring — Remote monitoring for patients with an ICD/CRT device

SUMMARY:
However, the current guidelines recommend the use of remote monitoring (RM) in patients with cardiac implantable electronic devices (CIED) to reduce inappropriate shocks or early detection of atrial fibrillation, data is incomprehensive on the effectiveness of decreasing heart failure events or mortality in patients with heart failure and reduced ejection fraction (HFrEF). The only randomized trial, which proved the efficacy of RM on mortality was the IN-TIME trial, which used a strict protocol for detection and intervention of the heart failure events.

The primary aim of this study is to optimize the use of remote monitoring system in HFrEF patients already implanted an implantable cardiac defibrillator (ICD) or a cardiac resynchronization therapy (CRT). By creating a high-quality system with structured safety-net, which is able to use the data of remote monitoring messages and alerts of our patients, we can improve their outcome. The primary endpoint is the non-fatal heart failure event or all-cause mortality. Secondary outcomes include all-cause mortality, cardiovascular mortality, heart failure hospitalization, cardiovascular hospitalization, unscheduled visits, af burden, stroke, inappropriate shocks, quality of life, NYHA functional class.

By using artificial intelligence-based methods, the optimal cut-off values of the previously, empirically used alert parameters will be validated or challenged. Additionally, cost-effectiveness to reduce the hospitalizations will be calculated.

Due to this remote monitoring structured safety-net, these patients with severe heart failure can be treated more efficiently, safely and cost-effectively.

ELIGIBILITY:
Inclusion Criteria:

1. CRT-P/CRT-D patients with a feasible device for home monitoring
2. ICD (VVI/VDD/DDD) patients with a feasible device for home monitoring
3. SR/AFib
4. Transmission performance >80% in the first 2 weeks with new device
5. Informed consent

Exclusion Criteria:

1. Life expectancy<1 year
2. Unable to transmit data
3. Patient is unable to visit the physician/clinic in 12 hours when it is indicated by the alerts
4. Expected non-compliance
5. Pregnancy
6. Known drug, alcohol abuse
7. Participation in other study or HM system concept

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic heart failure with reduced ejection fraction (HFrEF) with an implanted CIED (CRT/ICD) eligible for home monitoring
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The composite of all-cause mortality, heart failure events | 12 months

SECONDARY OUTCOMES:
cardiovascular mortality | 12 months
cardiovascular hospitalization | 12 months
unscheduled visits | 12 months

OTHER OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire score | 12 months
change of symptoms (assessed by NYHA classification) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University - Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes